CLINICAL TRIAL: NCT02241681
Title: Medium Chain Triglycerides Plasma Profile and Their Metabolites After Oral Peptamen Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14.22.MET
Record Dates: First submitted 2014-09-05; First posted 2014-09-16 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Medium Chain Triglycerides; Medium Chain Triglycerides metabolites; Peptamen 1.5

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peptamen 1.5 (Other): 500 mL of Peptamen 1.5
  Interventions: Dietary Supplement: Peptamen 1.5

INTERVENTIONS:
Dietary Supplement: Peptamen 1.5 — Peptamen will be given twice at the dose of 250 mL, with an interval of 4 hours.

SUMMARY:
Medium Chain Triglycerides (MCT) have been used for many years as a good source of lipid to decrease potential for fat malabsorption. However, the pharmacokinetics of MCT and of their metabolites have not been explored in details.

This is an exploratory study aiming at determining the plasma level of MCT and their metabolites after oral intake of Peptamen.

DETAILED DESCRIPTION:
20 subjects will be given 250mL of peptamen 1.5 twice, with 4 hours of interval, on a single day.

Plasma kinetics of MCTs and their metabolites will be made over 8 hours from baseline

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Aged between 20 and 65 years old
* BMI in the normal range (18.5 to 25.0 kg/m2)
* Having signed his/her consent form

Exclusion Criteria:

* Clinically relevant digestive (including malabsorption or major surgery), renal, hepatic, pancreatic or metabolic disease (diabetes, hypo or hyperthyroidism, hypo or hypercorticism), as determined by the medical (screening) visit and a standard blood chemistry analysis (glucose, total cholesterol, ALDL, AHDL, triglycerides, ASAT, ALTI, gamma GT, RCRP, creatinine)
* Medically diagnosed anemia based on a blood formula
* Food allergy, lactose intolerance and intolerance to milk proteins (anamnesis)
* Smokers (anamnesis)
* Pregnancy (anamnesis)
* Under corticoids or hormone (adrenal, thyroid) treatment
* Alcohol intake: > 2 units a day (anamnesis)
* Consumption of illicit drugs (anamnesis)
* Having given blood within the last month, or willing to make a blood donation until one month following the end of the study
* Subject who cannot be expected to comply with the study procedures, including consuming the test product
* Currently participating or having participated in another clinical trial during the last month prior to the beginning of this study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Measure of plasma Medium Chain Triglycerides (MCT) | over 8 hours post intake
  Tmax, Cmax and AUC for MCTs as compared to baseline.

SECONDARY OUTCOMES:
Measure of plasma MCT metabolites such as free fatty acids | over 8 hours post intake
  Tmax, Cmax and AUC for MCT metabolites as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD,PhD, Principal Investigator — Metabolic Unit, Clinical Development Unit,Nestec
Locations (1):
- Metabolic unit, clinical Development unit, Nestec, Lausanne, Switzerland